CLINICAL TRIAL: NCT04911361
Title: The DEPOT Study (Dry Eye Prescription Options for Therapy): A Randomized Controlled Clinical Trial Assessing the Efficacy and Safety of DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert, When Placed Within the Lower Eye Eyelid Canaliculus in Comparison to Topical Loteprednol Suspension for the Treatment of Episodic Dry Eye
Brief Title: The DEPOT Study (Dry Eye Prescription Options for Therapy)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEPOT 1911 OTX
Record Dates: First submitted 2021-04-02; First posted 2021-06-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized controlled, open label study of the efficacy of relieving both signs and symptoms of dry eye syndrome in patients with exacerbations of this disease. Patients will be randomized to receive treatment of either Dextenza or loteprednol etabonate 0.5% suspension QID for 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical loteprednol suspension in both eyes (Active Comparator): 25 subjects will be randomized to receive treatment loteprednol etabonate 0.5% suspension QID for 2 weeks.
  Interventions: Drug: Dexamethasone
- Lower eyelid canaliculi DEXTENZA insertion (study group) (Experimental): 25 subjects will be randomized to receive treatment of OTX-DED
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Patients will be randomized for either topical loteprednol suspension in both eyes (control group) or lower eyelid canaliculi DEXTENZA insertion (study group)
  Other Names: DEXTENZA

SUMMARY:
Assessing DEXTENZA efficacy and safety when placed within the lower eyelid canaliculus for dry eye flares in comparison to topical loteprednol suspension.

DETAILED DESCRIPTION:
The DEPOT Study (Dry Eye Prescription Options for Therapy): A randomized controlled clinical trial assessing the efficacy and safety of DEXTENZA, sustained release dexamethasone 0.4 mg insert, when placed within the lower eye eyelid canaliculus in comparison to topical loteprednol suspension for the treatment of episodic dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Patients willing to take an electronic survey about their tolerability of either study medication.
* Patients with a recent exacerbation of dry eye characterized by ocular surface discomfort.

Exclusion Criteria:

* Active, systemic or local disease condition other than DES that causes clinically significant ocular surface irritation that could interfere with the evaluation and treatment of dry eye.
* Any of the following ocular (eye or eyelid) conditions in either eye within 1 Months prior to the enrollment visit:

  * Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgery procedure)
  * Clinically significant ocular trauma.
  * Active ocular Herpes simplex or Herpes zoster (eye or eyelid) infection.
  * Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis)
  * Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye)
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis
* Eyelid abnormalities that significantly affect lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis)
* Ocular surface abnormality that may compromise corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy)
* Participation in another ophthalmic clinical trial involving a therapeutic drug or device within 30 days prior to the distribution of the survey
* Participation in this trial in the same patient's fellow eye.
* Patients who are pregnant or breastfeeding or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
To determine effect of dexamethasone insert | 2 Weeks
  SPEED score at Baseline and Week 2

SECONDARY OUTCOMES:
To determine the effect of dexamethasone insert | 4 Weeks
  The difference in SPEED questionnaire scores before and 4 weeks after treatment.
The difference in conjunctival hyperemia | 4 weeks
  Slit exam to determine ocular hyperemia using the Schulze Scale before and 4 weeks after treatment
The difference in tear break up time (TBUT) before and after treatment | 4 Weeks
  Reduced tear break up time (TBUT) ≤ 10 seconds
The difference in corneal staining before and after treament | 4 Weeks
  The presence of central or inferior staining defined by the Oxford Scale

OTHER OUTCOMES:
Safety outcome measure | At baseline, 2 weeks, and 4 weeks
  Intraocular pressure at Baseline, Week 2 & 4

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Research Insight LLC
Locations (3):
- United States (3):
  - Inland Eye Specialists, Hemet, California
  - Harvard Eye Associates, Laguna Hills, California
  - Ophthalmology Associates, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
IPD results will be shared in publication.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938
- [Background] Walters TR, et al. Efficacy and Safety of Sustained Release Dexamethasone for the Treatment of Ocular Pain and Inflammation after Cataract Surgery: Results from Two Phase 3 Studies. J Clin Exp Ophthalmol. 2016; 7(4):
- See also: DEXTENZA (dexamethasone insert) Prescribing Information, Ocular Therapeutix,Inc.2019 — http://www.dextenza.com/wp-content/uploads/2019/06/NDA-208742-S001-Dextenza-labeling-19Jun19.pdf